CLINICAL TRIAL: NCT02304783
Title: The Investigation of the Efficacity and Safety of Oral Non Steroidal Anti Inflammatory (NSAI) Drugs Such as Piroxicam as a Second Line Treatment of Patients Consulting the Emergency Departement for Renal Colics.
Brief Title: Oral NSAI Versus Paracetamol or Placebo as a Second Line Treatment for Renal Colics
Acronym: ONSAIP-RC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Oral NSAI in RC
Record Dates: First submitted 2014-11-26; First posted 2014-12-02 (Estimated); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Renal Colic
Keywords: Renal colic, Piroxicam
MeSH Terms: conditions — Renal Colic | interventions — Piroxicam; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oral Piroxicam (Active Comparator): Piroxicam : 20 mg per pill; one pill per day for five days associated with placebo (1pill) (taken separately)
  Interventions: Drug: Piroxicam
- Placebo (Placebo Comparator): Placebo: two pills per day for five days (taken separately)
  Interventions: Drug: Placebo
- paracetamol (Active Comparator): paracetamol: 2000mg per day for five days two pills taken separately)
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: Piroxicam — Patients allocated to this arm received, as a second line treatment of renal colics, a five days treatment with 20 mg piroxicam associated with placebo per day and were contacted at the seventh day by telephone call to investigate the efficacity and the side effects of the treatment.
  Other Names: Piroxen
  Arms: Oral Piroxicam
Drug: Placebo — Patients allocated to this arm received a five days treatment with Placebo and were contacted at the seventh day by telephone call to investigate the efficacity and the side effects of the treatment.
  Arms: Placebo
Drug: paracetamol — Patients allocated to this arm received a five days treatment with Paracetamol and were contacted at the seventh day by telephone call to investigate the efficacity and the side effects of the treatment.
  Arms: paracetamol

SUMMARY:
Outpatients treatment with NSAI in renal colics has not been well investigated and there is no clear recommendations regarding this matter.

The aim of this study is to determine if an oral NSAI treatment is beneficial in patients discharged for the emergency departement after the first line treatment of a renal colic investigating the recurrence of pain, the reconsultation rates and the admissions.

DETAILED DESCRIPTION:
Renal colic (RC)are a frequent cause of consultation in the emergency departement (ED).

They count for approximatively 20% of patients presenting to the ED with severe acute onset abdominal pain.

The first line treatment of renal colics is based on NSAI drugs associated with antalgics and is further investigated in the NSAI vs Morphine study (NCT02156596).

But there is no clear recommendations regarding the outpatient treatment of renal colics.

Oral NSAI are still widely used as a second line medicine for this condition and variety of molecules were tried with no solid scientific arguments.

Piroxicam, a non-selective COX inhibitor drug appared to the Oxicam class of NSAI, is widely used to treat rheumatoid conditions and other inflammatory conditions and often prescribed in Tunisia as a second line treatment of RC.

In this study, we aimed to investigate the efficiency and safety of the use of oral NSAI drugs (Piroxicam) compared to paracetamol or placebo as a second line treatment of renal colics.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Consenting to participate in the study
* Patients treated in the ED for RC
* No contraindications of NSAI treatment

Exclusion Criteria:

* Patients excluded from the first phase of the study
* Contraindication of NSAI treatment
* Patients non reachable by telephone call
* Patients that did not receive or use the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Efficacity of oral NSAI (telephone call, asking for the recurrence of pain, the reconsultation rates and intervals and the need for other treatments) | seven days
  The efficacity of the oral NSAI treatment was evaluated at the seventh day by a telephone call, asking for the recurrence of painand the readmission rates)

SECONDARY OUTCOMES:
Safety of NSAI (telephone call, asking for mean time to recurrence and the occurence of NSAI side effects such as abdominal pain, vomiting, rush, bleeding and ect) | seven days
  The efficacity of the oral NSAI treatment was evaluated at the seventh day by a telephone call, asking for the occurence of NSAI side effects such as abdominal pain, vomiting, rush, bleeding and ect

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, MD, Principal Investigator — University of Monastir
Locations (1):
- Emergency Department of University Hospital of Monastir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: official department site — http://www.urgencemonastir.com